CLINICAL TRIAL: NCT05886452
Title: Success of Dailies Total1 for Astigmatism Contact Lenses in Patients That Have Previously Failed With Toric Contact Lenses
Status: Completed | Type: Observational
Sponsor: Mann Eye Institute (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: PB-23-02
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- DT1fA contact lenses: Subjects fitted with DT1fA contact lenses
  Interventions: Device: DT1fA contact lenses

INTERVENTIONS:
Device: DT1fA contact lenses — Subjects will be fitted with DT1fA contact lenses

SUMMARY:
The objective is to determine the percentages of past toric CL wearers (who dropped out of contact lens wear due to dissatisfaction with comfort or vision) who are satisfied with the comfort and vision of DT1fA contact lenses.

DETAILED DESCRIPTION:
This is a single arm, prospective, non-comparative, open-label post market clinical study of satisfaction of past toric CL wearers, with DT1fA contact lenses. Subjects will be assessed at a screening visit, and 2 follow-up visits. Clinical evaluations will include measurement of visual acuity, manifest refraction, and administration a questionnaire

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

* Gender: Males and Females.
* Subjects will be 18-39 years old.
* History of previous unsuccessful astigmatism contact lens wearer with qualifying answer to screening questions:

  * I used to wear astigmatism correcting (toric) soft contact lenses.

    - (YES)
  * I stopped wearing my previous astigmatism correcting soft contact lenses because of one or more of the below reasons:

    * Poor or fluctuating vision
    * Discomfort
    * Other
* Subjects must have 20/25 or better distance visual acuity in each eye with current best correction.
* Good general health (defined by prescription medication use that has not changed within the last month and the absence of medical conditions or treatments that are deemed confounding to the data as determined by the PI).
* Ability to give informed consent.
* Willing and able to spend time for the study (Subjects will be required to attend three study visits and wear contact lenses on days between study visits).

Exclusion Criteria:

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Previous ocular surgery.
* Inability to be fit with the DT1fA lens design.
* Subjects that should be wearing a toric contact lens for best acuity but have chosen to continue in spherical contact lens wear.
* History of Accutane use.
* Ocular surface disease that in the investigator's opinion would interfere with contact lens wear.
* History of comorbidities, including autoimmune disorders and diabetes.
* Irregular astigmatism as identified by Pentacam.
* History of Amblyopia.
* History of Strabismus and/or history of eye muscle surgery.
* History of Monovision.
* Potential subjects who are pregnant.

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Ages: 18 Years to 39 Years | Sex: All
Age Groups: Adult
Study Population: Eligible test subjects will be 18 to 39 years of age with history of previous unsuccessful astigmatism contact lens wear.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Brunson, OD, Principal Investigator — Mann Eye Institute
Locations (1):
- Mann Eye Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DT1fA Contact Lenses
Started | 65
Completed | 65
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | DT1fA Contact Lenses
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Positive Ratings (>50 Out of 100) for Satisfaction of Comfort and Vision.
Description: A questionnaire will be administered. Subjects are asked to rate their satisfaction with comfort and vision on a scale of 0 to 100, with higher ratings indicating higher satisfaction with comfort and vision.
Time Frame: After 30 days of DT1fA contact lens wear
Measure: Count of Participants; unit: Participants
Arm/Group | DT1fA Contact Lenses
Number analyzed (Participants) | 65
Participants | 57

2. Other Pre Specified Outcome: Percentage of Patients Reporting Satisfaction of Overall and End of Day (EOD) Comfort and Vision; Comfort and Vision Under Real-world Conditions Related to Computer (or Tablet) Usage and Cellphone Usage.
Description: A questionnaire will be administered. Subjects are asked to rate their satisfaction with end of day comfort and vision on a Likert scale (Strongly Disagree, Disagree, Neither Disagree nor Agree, Agree, Strongly Agree). Satisfaction was determined as subjects answering "Agree" or "Strongly Agree".
Time Frame: After 30 days of DT1fA contact lens wear
Measure: Count of Participants; unit: Participants
Arm/Group | DT1fA Contact Lenses
Number analyzed (Participants) | 65
Participants | 36

3. Other Pre Specified Outcome: Percentage of Patients Reporting a Desire to Remain in DT1fA Lenses After Study is Concluded.
Description: A questionnaire will be administered. Subjects are asked to rate their desire to remain in DT1fA contact lenses a Likert scale (Strongly Disagree, Disagree, Neither Disagree nor Agree, Agree, Strongly Agree). Desire to remain was determined as subjects answering "Agree" or "Strongly Agree".
Time Frame: After 30 days of DT1fA contact lens wear
Measure: Count of Participants; unit: Participants
Arm/Group | DT1fA Contact Lenses
Number analyzed (Participants) | 65
Participants | 38

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | DT1fA Contact Lenses
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT05886452/Prot_SAP_000.pdf